CLINICAL TRIAL: NCT04606667
Title: Multicomponent Exercise in the Functionality of the Elderly in the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Piaget (Other)
Responsible Party: Principal Investigator, José Luís Alves Sousa, Physiotherapy coordinator, Instituto Piaget
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: InstitutoPiaget
Record Dates: First submitted 2020-09-18; First posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Aging; Cognition; Balance; Mobility Limitation
Keywords: Aging; Community; Exercise program; Physiotherapy; Functionality
MeSH Terms: conditions — Mobility Limitation | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Quasi-experimental, test-retest, with one sample.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multi component program (Experimental): The intervention lasted 16 weeks, with the evaluations carried out at baseline, after 8 weeks and at the end.
  The multi-component exercise program took place in day centers or collective residences. It was supervised by physiotherapists. The classes took place 3 times a week, at the same hour and on alternate days, for 45-60 minutes, for a total of 48 sessions. The program consisted on a warm-up (5 min) with exercises and walking, a balance and strength training (35-40 min) with exercises repeated 3 times and held for 15 seconds flexibility / relaxation (5 to 10 mins) periods. The strength training is performed with the resistance of the body weight or accessible and low cost equipment, with two series of 10 to 15 repetitions, after maximum resistance was calculated.
  The flexibility and cooling training consists of 3 repetitions maintained for 15 seconds.
  Interventions: Other: Exercise Program

INTERVENTIONS:
Other: Exercise Program — Exercise program

SUMMARY:
Evaluate the results of the implementation of a multicomponent exercise program (16 weeks) for elder community dwelling population on their functionality (via cognitive, balance and mobility status).

DETAILED DESCRIPTION:
A quasi-experimental study, of the pre-test-post-test type, with a sample for convenience from in a cohort of elderly community dwelling people, carried out between 2009 and 2011. The general objective is to verify the impact of a physical exercise program organized in classes, under the supervision of physiotherapists.The specific objectives are to analyze the effect after 8 and 16 weeks, on the functionality of the elderly person, discriminating three conditions: cognitive state, balance and functional mobility.

ELIGIBILITY:
Inclusion Criteria:

* be supported by day centers or collective residences linked to the "Project + City",
* not having regular exercise habits,
* ability to walk (with or without assistance).

Exclusion Criteria:

* not being collaborative,
* missing the classes three times.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Functional mobility change | Baseline, 8 weeks, 16 weeks
  Timed Up and Go Test is a validated test that consists on a timed 3 meter defined circuit after getting up from a chair and sitting in it. The categories of achievement are three: less than 10 seconds "without compromise", corresponding to normal performance; between 10.01 and 20 seconds it is considered "slight impairment or normal time for frail elderly"; more than 20.01 seconds corresponds to a degree of "functional impairment" that requires a more detailed assessment.
Balance change | Baseline, 8 weeks, 16 weeks
  Berg scale is a validated instrument to assess balance and the risk of falling associated with its loss. From 56 to 54 points, each point less is associated with a 3 to 4% increase in the risk of falling, from 54 to 46 a change in one point is associated with a 6 to 8% increase in the risk of falling, and below 36 points the risk of falling is very close to 100%, which allows the results to be divided into 4 balance categories: "Total balance problem" (≤36 points); "Serious balance problem" (37-45 points); "Moderate balance problem" (46-53 points) and "normal balance" (≥54 points).
Cognitive status change | Baseline, 8 weeks, 16 weeks
  Mini mental exam scale is a validate instrument to assess the cognitive function and the detection of potential dementia. Individuals are classified into three categories: a score equal to or less than 18 points corresponds to "severe cognitive impairment"; from 19 to 23 points "moderate cognitive impairment" and 24 or more points "normal cognitive state. The literature states that for the diagnosis of dementia, the scale results must be cross-checked with schooling, however when the objective is not to diagnose dementia, but only to characterize and assess changes in cognitive status, the crossing of the scale results with schooling does not justified.

CONTACTS AND LOCATIONS:
Overall Officials: José LA Sousa, PhD, Principal Investigator — Instituto Piaget
Locations (1):
- Escola Superior de Saúde, Vila Nova de Gaia, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American College of Sports Medicine; Chodzko-Zajko WJ, Proctor DN, Fiatarone Singh MA, Minson CT, Nigg CR, Salem GJ, Skinner JS. American College of Sports Medicine position stand. Exercise and physical activity for older adults. Med Sci Sports Exerc. 2009 Jul;41(7):1510-30. doi: 10.1249/MSS.0b013e3181a0c95c. PMID 19516148
- [Background] Boyle PA, Buchman AS, Wilson RS, Bienias JL, Bennett DA. Physical activity is associated with incident disability in community-based older persons. J Am Geriatr Soc. 2007 Feb;55(2):195-201. doi: 10.1111/j.1532-5415.2007.01038.x. PMID 17302655
- [Background] Cadore EL, Rodriguez-Manas L, Sinclair A, Izquierdo M. Effects of different exercise interventions on risk of falls, gait ability, and balance in physically frail older adults: a systematic review. Rejuvenation Res. 2013 Apr;16(2):105-14. doi: 10.1089/rej.2012.1397. PMID 23327448
- [Background] Gine-Garriga M, Roque-Figuls M, Coll-Planas L, Sitja-Rabert M, Salva A. Physical exercise interventions for improving performance-based measures of physical function in community-dwelling, frail older adults: a systematic review and meta-analysis. Arch Phys Med Rehabil. 2014 Apr;95(4):753-769.e3. doi: 10.1016/j.apmr.2013.11.007. Epub 2013 Nov 27. PMID 24291597
- [Background] Gschwind YJ, Kressig RW, Lacroix A, Muehlbauer T, Pfenninger B, Granacher U. A best practice fall prevention exercise program to improve balance, strength / power, and psychosocial health in older adults: study protocol for a randomized controlled trial. BMC Geriatr. 2013 Oct 9;13:105. doi: 10.1186/1471-2318-13-105. PMID 24106864
- [Background] Sjosten NM, Salonoja M, Piirtola M, Vahlberg T, Isoaho R, Hyttinen H, Aarnio P, Kivela SL. A multifactorial fall prevention programme in home-dwelling elderly people: a randomized-controlled trial. Public Health. 2007 Apr;121(4):308-18. doi: 10.1016/j.puhe.2006.09.018. Epub 2007 Feb 22. PMID 17320125
- [Background] Lee HC, Chang KC, Tsauo JY, Hung JW, Huang YC, Lin SI; Fall Prevention Initiatives in Taiwan (FPIT) Investigators. Effects of a multifactorial fall prevention program on fall incidence and physical function in community-dwelling older adults with risk of falls. Arch Phys Med Rehabil. 2013 Apr;94(4):606-15, 615.e1. doi: 10.1016/j.apmr.2012.11.037. Epub 2012 Dec 6. PMID 23220343
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Guerreiro, MPSA, et al. Adaptação à população portuguesa da tradução do Mini Mental State Examination (MMSE). Revista Portuguesa de Neurologia, 1994, 1.9: 9-10.
- [Background] Berg KO, Wood-Dauphinee SL, Williams JI, Maki B. Measuring balance in the elderly: validation of an instrument. Can J Public Health. 1992 Jul-Aug;83 Suppl 2:S7-11. PMID 1468055
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Shumway-Cook A, Baldwin M, Polissar NL, Gruber W. Predicting the probability for falls in community-dwelling older adults. Phys Ther. 1997 Aug;77(8):812-9. doi: 10.1093/ptj/77.8.812. PMID 9256869
- [Background] Bherer L, Erickson KI, Liu-Ambrose T. A review of the effects of physical activity and exercise on cognitive and brain functions in older adults. J Aging Res. 2013;2013:657508. doi: 10.1155/2013/657508. Epub 2013 Sep 11. PMID 24102028
- [Background] Freiberger E, Menz HB, Abu-Omar K, Rutten A. Preventing falls in physically active community-dwelling older people: a comparison of two intervention techniques. Gerontology. 2007;53(5):298-305. doi: 10.1159/000103256. Epub 2007 May 29. PMID 17536207